CLINICAL TRIAL: NCT00242411
Title: A Comparison of the Efficacy of Symbicort® Single Inhaler Therapy (Symbicort Turbuhaler® 160/4.5 mg 1 Inhalation b.i.d. Plus As-needed) and Conventional Best Standard Treatment for the Treatment of Persistent Asthma in Adolescents and Adults. A Randomized, Open, Parallel-group, Multicentre 26-weeks Study
Brief Title: MONO: Symbicort® Single Inhaler Therapy and Conventional Best Standard Treatment for the Treatment of Persistent Asthma in Adolescents and Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5890L00008
Record Dates: First submitted 2005-10-18; First posted 2005-10-20 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

INTERVENTIONS:
Drug: Budesonide/Formoterol Turbuhaler
Drug: Conventional Best Asthma Therapy

SUMMARY:
The purpose of the study is to compare the efficacy of a flexible dose of Symbicort (budesonide/formoterol) with conventional stepwise best standard treatment in patients with persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma >= 3 months
* Prescribed daily use of glucocorticosteroids for at least 3 months prior to Visit 1

Exclusion Criteria:

* Smoking history > 10 pack-years
* Asthma exacerbation requiring change in asthma treatment during the last 14 days prior to inclusion
* Any significant disease or disorder that may jeopardize the safety of the patient.

Additional inclusion and exclusion criteria will be evaluated by the investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1900
Dates: Start 2004-09; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Time to first severe asthma exacerbation

SECONDARY OUTCOMES:
Number of asthma exacerbations
Mean use of as-needed medication
Prescribed asthma medication
Asthma Control Questionnaire
Safety: serious adverse events and discontinuations due to adverse events
All variables assessed over the 6 month treatment period

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Symbicort Medical Science Director, MD, Study Director — AstraZeneca
Locations (179):
- Denmark (86):
  - Research Site, Aabenraa
  - Research Site, Aalborg
  - Research Site, Albertslund
  - Research Site, Allingåbro
  - Research Site, Ålbæk
  - Research Site, Ålestrup
  - Research Site, Århus C
  - Research Site, Bagsværd
  - Research Site, Ballerup Municipality
  - Research Site, Billund
  - Research Site, Birkerød
  - Research Site, Brønderslev
  - Research Site, Brønshøj
  - Research Site, Ejby
  - Research Site, Fåborg
  - Research Site, Fredericia
  - Research Site, Frederiksberg
  - Research Site, Frederiksberg C
  - Research Site, Frederikshavn
  - Research Site, Frederikssund
  - Research Site, Glesborg
  - Research Site, Glumsø
  - Research Site, Greve
  - Research Site, Hårlev
  - Research Site, Hellerup
  - Research Site, Helsinge
  - Research Site, Herning
  - Research Site, Hillerød
  - Research Site, Holbæk
  - Research Site, Hornbæk
  - Research Site, Horsens
  - Research Site, Humlebæk
  - Research Site, Hvidovre
  - Research Site, Ikast
  - Research Site, Jægerspris
  - Research Site, Karlslunde
  - Research Site, Kåstrup
  - Research Site, Kjellerup
  - Research Site, Klarup
  - Research Site, Kolding
  - Research Site, Kolind
  - Research Site, Korsør
  - Research Site, Kværndrup
  - Research Site, København K
  - Research Site, København S
  - Research Site, København Ø
  - Research Site, Lynge
  - Research Site, Lystrup
  - Research Site, Nakskov
  - Research Site, Nibe
  - Research Site, Nyborg
  - Research Site, Nykøbing Falster
  - Research Site, Nærum
  - Research Site, Næstved
  - Research Site, Nørre Alslev
  - Research Site, Nørresundby
  - Research Site, Odense C
  - Research Site, Odense NV
  - Research Site, Oksbøl
  - Research Site, Randers
  - Research Site, Redsted
  - Research Site, Ringsted
  - Research Site, Risskov
  - Research Site, Roskilde
  - Research Site, Rudkøbing
  - Research Site, Rungsted Kyst
  - Research Site, Rødovre Municipality
  - Research Site, Saltum
  - Research Site, Skibby
  - Research Site, Slagelse
  - Research Site, Stensved
  - Research Site, Struer Municipality
  - Research Site, Sulsted
  - Research Site, Svendborg
  - Research Site, Sæby
  - Research Site, Sønderborg
  - Research Site, Søndersø
  - Research Site, Tåstrup
  - Research Site, Thorsø
  - Research Site, Tølløse
  - Research Site, Tønder
  - Research Site, Varde
  - Research Site, Viborg
  - Research Site, Viby J
  - Research Site, Vojens
  - Research Site, Ølstykke
- Finland (42):
  - Research Site, Anjalankoski
  - Research Site, Espoo
  - Research Site, Hammaslahti
  - Research Site, Harjavalta
  - Research Site, Heinola
  - Research Site, Helsingin Kaup
  - Research Site, Helsinki
  - Research Site, Jakobstad
  - Research Site, Joensuu
  - Research Site, Joutseno
  - Research Site, Jyväskylä
  - Research Site, Kajaani
  - Research Site, Kinkomaa
  - Research Site, Kotka
  - Research Site, Kouvola
  - Research Site, Kuusamo
  - Research Site, Lahti
  - Research Site, Lappeenranta
  - Research Site, Lapua
  - Research Site, Lieto
  - Research Site, Lohja
  - Research Site, Mäntsälä
  - Research Site, Mikkeli
  - Research Site, Muhos
  - Research Site, Nokia
  - Research Site, Oulu
  - Research Site, Parkano
  - Research Site, Pattijoki
  - Research Site, Polvijärvi
  - Research Site, Pori
  - Research Site, Porvoo
  - Research Site, Ristiina
  - Research Site, Rovaniemi
  - Research Site, Savonlinna
  - Research Site, Tampere
  - Research Site, Tornio
  - Research Site, Turku
  - Research Site, Vantaa
  - Research Site, Varkaus
  - Research Site, Vimpeli
  - Research Site, Ylitornio
  - Research Site, Ylöjärvi
- Norway (51):
  - Research Site, Aksdal
  - Research Site, Arendal
  - Research Site, Asker
  - Research Site, Årnes
  - Research Site, Bergen
  - Research Site, Bodø
  - Research Site, Drammen
  - Research Site, Fevik
  - Research Site, Fjerdingby
  - Research Site, Flatåsen
  - Research Site, Fredrikstad
  - Research Site, Fyllingsdalen
  - Research Site, Hafrsfjord
  - Research Site, Harstad
  - Research Site, Haugesund
  - Research Site, Hosle
  - Research Site, Høvik
  - Research Site, Karmsund
  - Research Site, Kristiansand
  - Research Site, Lena
  - Research Site, Lier
  - Research Site, Lierskogen
  - Research Site, Lillestrøm
  - Research Site, Lysaker
  - Research Site, Lørenskog
  - Research Site, Løvenstad
  - Research Site, Molde
  - Research Site, Nesbru
  - Research Site, Nesttun
  - Research Site, Oslo
  - Research Site, Paradis
  - Research Site, Rådal
  - Research Site, Rykkin
  - Research Site, Røa
  - Research Site, Sandvika
  - Research Site, Skedsmokorset
  - Research Site, Ski
  - Research Site, Skien
  - Research Site, Slependen
  - Research Site, Spikkestad
  - Research Site, Steinkjer
  - Research Site, Straume
  - Research Site, Strømmen
  - Research Site, Svelvik
  - Research Site, Søgne
  - Research Site, Sørumsand
  - Research Site, Tolvsrød
  - Research Site, Trollåsen
  - Research Site, Tromsø
  - Research Site, Trondheim
  - Research Site, Ulset